CLINICAL TRIAL: NCT00222833
Title: The Effect of Switching to Aripiprazole on Indices of Cardiovascular Health in Overweight and Obese Patients With Schizophrenia
Brief Title: The Effect of Switching to Aripiprazole on Heart Health in Overweight and Obese Patients With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0312010; PITT#02 90599
Record Dates: First submitted 2005-09-07; First posted 2005-09-22 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2008-01

CONDITIONS: Overweight; Hyperlipidemia; Cardiovascular Diseases
Keywords: Schizophrenia; Schizoaffective disorder; Aripiprazole; Obese; Overweight; Heart Health; Antipsychotic; Heart Health Factors; Cardiovascular Health Indices; Cardiovascular health
MeSH Terms: conditions — Overweight; Hyperlipidemias; Cardiovascular Diseases; Schizophrenia; Psychotic Disorders; Obesity | interventions — Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole

SUMMARY:
This is a 2-year study proposing to examine the effects of aripiprazole on heart health factors such as serum lipids, serum leptin, fasting blood sugar, body weight and blood pressure. This study also examines the safety of switching to aripiprazole with respect to changes in the clinical state, preexisting or emergent side-effects, how the brain processes information and changes in social functioning and quality of life.

DETAILED DESCRIPTION:
This is a 2-yr study proposing to examine the effects of switching subjects from conventional and atypical antipsychotic agents to Aripiprazole on cardiovascular health indices in overweight and obese patients with Schizophrenia or Schizoaffective disorder. Thirty partially remitted patients with Positive and Negative Syndrome Scale (PANSS) score of less than 100, who have body mass index (BMI) of 26 or higher will be switched from their existing antipsychotic to aripiprazole over 2-3 weeks period using a clinician determined cross-tapering approach.The objective of the study is to examine cardiovascular health indices such as serum lipids, serum leptin, fasting blood sugar, body weight and blood pressure. This study also examines the safety of switching to Aripiprazole with respect to changes in clinical state, preexisting or emergent side-effects, how brain processes information and changes in social functioning and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ages 18-65 years
* Outpatients and stable partial hospital patients
* Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) diagnosis of schizophrenia or schizoaffective disorder
* No psychiatric hospitalization in 30 days prior to study start
* Partially remitted patients with a PANSS score below 100 at screening
* Currently on a stable dose of only one antipsychotic for at least 30 days prior to study start
* Currently receiving a stable dose of all other psychotropic medications for at least 30 days prior to study start
* BMI greater than 26
* Female patients of childbearing age must be using an acceptable method of birth control for at least 1 month prior to participation in the research study and continue for at least 4 weeks after the final study visit.
* Ability to provide informed consent.

Exclusion Criteria:

* Mental retardation
* Current treatment with clozapine
* Currently enrolled in a weight management program or receiving pharmacological treatment for weight reduction
* Serious or unstable medical illness
* Female patients who are pregnant, lactating, or plan to become pregnant during the study period
* Concurrently receiving treatment with ketoconazole, quinidine, carbamazepine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-10; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
To examine heart health factors: serum lipids, serum leptin, fasting blood glucose, body weight, and blood pressure

SECONDARY OUTCOMES:
Changes in clinical state
Pre-existing or emergent side effects
Cognition and insight
Attitude towards medication
Social functioning
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Rohan Ganguli, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Institute and Clinic of UPMC, Pittsburgh, Pennsylvania, United States